CLINICAL TRIAL: NCT05332782
Title: Outcomes of Patients tReated wIth Mitral Transcatheter Edge-to-edge Repair for Primary Mitral Regurgitation Registry
Acronym: PRIME-MR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PRIME-MR
Record Dates: First submitted 2022-03-01; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- M-TEER: Patients with primary mitral regurgitation undergoing mitral valve transcatheter edge-to-edge repair.

SUMMARY:
This multinational, non-interventional, investigator-initiated, retrospective study aims to investigate outcomes of patients, who underwent mitral valve transcatheter edge-to-edge repair (M-TEER) for primary mitral regurgitation (PMR).

ELIGIBILITY:
Inclusion Criteria:

* clinically significant primary mitral regurgitation
* patient underwent M-TEER
* echocardiography data at baseline, procedure and follow-up
* follow-up of at least 12 months

Exclusion Criteria

* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing transcatheter edge-to-edge repair for primary mitral regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 months
  Incidence of death from any cause.
Cardiovascular mortality | 12 months
  Incidence of cardiovascular death, defined as death attributable to myocardial ischemia and infarction, heart failure, cardiac arrest because of other or unknown cause, or cerebrovascular accident.
Rehospitalization for congestive heart failure | 12 months
  Incidence of new-onset or worsening signs and symptoms of heart failure that required urgent therapy and resulted in hospitalization, e.g. as assessed by patient interviews or medical records.
Re-do mitral valve procedure | 12 months
  Incidence of unplanned surgical (mitral valve repair or replacement) or transcatheter re-intervention (re-do transcatheter edge-to-edge repair), e.g. as assessed by patient interviews or medical records.

SECONDARY OUTCOMES:
Residual mitral regurgitation | up to 30 days
  Mitral regurgitation severity (0, 1+, 2+, 3+, 4+) as assessed by transthoracic echocardiography at discharge.
Residual mitral regurgitation | 12 months
  Mitral regurgitation severity (0, 1+, 2+, 3+, 4+) as assessed by transthoracic echocardiography at 1-year follow-up.
MVARC (Mitral Valve Academic Research Consortium) Technical success | 1 day (at exit from the catheterization laboratory)
  All of the following must be present:
  1. Absence of procedural mortality
  2. Successful access, delivery, and retrieval
  3. Successful deployment and correct positioning of the first device
  4. Freedom from emergency surgery or reintervention related to the device or access procedure
Functional success | 1 day (at exit from the catheterization laboratory)
  If one of the following is present:
  1. Residual mitral regurgitation ≤2+
  2. Effective regurgitant orifice area ≤15 mm2
  3. Transmitral gradient <5 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kalbacher, MD, Principal Investigator — University Heart & Vascular Center Hamburg
Locations (6):
- Montefiore Medical Center, New York, New York, United States
- France (3):
  - Centre Hospitalier de Bordeaux, Bordeaux
  - Université Lille, Inserm, Centre Hospitalier Universitaire de Lille, Lille
  - University Hospital of Rennes, Centre Hospitalier de Rennes, Rennes
- Germany (2):
  - University Heart & Vascular Center Hamburg, Hamburg
  - Klinikum der Universität München, Munich

IPD SHARING:
Plan to Share IPD: No